CLINICAL TRIAL: NCT04248556
Title: Dermatological Assessment of Primary Dermal Irritability Accumulated and Sensitization Under Controlled and Maximised Conditions
Brief Title: Dermatological Assessment of Primary Dermal Irritability Accumulated and Sensitization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: All-S-RIPT-SO-PAD-074832
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Sensitivity, Contact
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Intervention Model Description: Clinical trial, single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subjects, 18-59 y, healthy (Experimental): patch test with investigation product
  Interventions: Other: Health care product

INTERVENTIONS:
Other: Health care product — Health care product (gel) - to be applied on the participant's skin

SUMMARY:
This is a clinical study for health care product safety assessment. The research will be conducted with 92 subjects, aged 18 to 59 years. The product will be applied on the right and/or left back of the research participants for 3 consecutive weeks. After 10 days, will have another application of the same product, which will be removed in 48 hours. Medical evaluation will be available throughout the study to assess possible adverse events.

The objective of the study is to observe the effects of the application of the product on the skin and prove the absence of irritability and/or allergy.

DETAILED DESCRIPTION:
92 subjects, aged 18 to 59 years, phototypes I to IV (according to Fitzpatrick classification). The patch test will be used to verify the absence of primary and cumulative dermal irritation reactions and sensitization allergic reactions by the investigational products. The products will be applied as they are over semi-occlusive dressings.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to comply with safety guidelines to minimize contamination risks to COVID-19;
* Agreement to perform a molecular test to detect COVID-19 to enter the study;
* Healthy participants;
* Non-injured skin in the test region;
* Agreement to adhere to the test procedures and requirements and to attend the institute on the day(s) and at the time(s) determined for the evaluations;
* ability to consent to participation in the study;
* Age from 18 to 59 years;
* Phototype (Fitzpatrick): I to IV;
* All sex.

Exclusion Criteria:

* Participants who belong to the risk group for COVID-19, that is, with diabetes, with chronic cardiovascular, renal and respiratory problems, immunosuppressed or other conditions that the doctor deems to belong to the risk group;
* Pregnant or breastfeeding women;
* Skin marks in the experimental area that interfere with the evaluation of possible skin reactions;
* Active dermatoses;
* Background of allergic reactions, irritation or intense discomfort sensations to topical use products;
* History of atopy (atopic dermatitis, allergic rhinitis, allergic bronchitis, allergic conjunctivitis, etc.);
* Sensation of discomfort with temperature changes (too hot/very cold) and/or when in the air conditioning;
* Participants with a history of allergy to materials used in the study;
* History of pathologies aggravated or triggered by ultraviolet radiation;
* Carriers of immunodeficiencies;
* Intense sun exposure or tanning session up to 15 days before the initial evaluation;
* Prediction of intense sun exposure or tanning session during the course of the study;
* Expected to bathe in the sea, pool or bathtub during the conduct of the study;
* Participants who practice water sports;
* Dermography;
* Aesthetic and/or body dermatological treatment until 03 weeks before the selection;
* Use of the following topical or systemic drugs: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs and corticoids until 2 weeks before selection or, considering deposit corticoids, the interval shall be 1 month before selection;
* Treatment with acidic vitamin A and/or its derivatives via oral or topical up to 1 month before the start of the study;
* Vaccination during the study or up to 3 weeks before the study;
* Being or having participated in another clinical trial terminated less than 7 days before selection, if the previous trial is acceptable in use;
* Being or having participated in another clinical trial terminated less than 21 days before the selection, in case the previous trial is compatible or Adverse Reaction investigative;
* Any condition not mentioned above that, in the opinion of the investigator, may compromise the assessment of the trial;
* History of no adherence or unwillingness to adhere to the study protocol;
* Professionals directly involved in the conduct of this protocol and their families.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
Absence | 4 weeks
  Absence of the occurrence of reactions of primary, accumulated dermal irritation and of allergic reactions by sensitization by the investigational products.

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, São Paulo, Brazil